CLINICAL TRIAL: NCT04509765
Title: A Phase II Single-Arm Study of Total Body Irradiation With Linac Based Volumetric Modulated Arc Therapy (VMAT) and Image Guided Radiation Therapy (IGRT)
Brief Title: A Phase II Single-arm Study of Total Body Irradiation With Linac Based VMAT and IGRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00664
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Malignancy
Keywords: Myeloablative Treatment; Total Body Irradiation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with Hematologic Malgnancies (Experimental)
  Interventions: Radiation: Linac Based VMAT TBI

INTERVENTIONS:
Radiation: Linac Based VMAT TBI — Use of linac based Volumetric Arc Therapy (VMAT) to deliver Total Body Irradiation (TBI). The study intervention is a VMAT based delivery technique using a 6 MV photon beam from a Varian TrueBeam® (Palo Alto, CA) equipped with a Millennium multi-leaf collimation (MLC) system3. TBI will be delivered using a Varian TrueBeam linear accelerator with photon beam VMAT capability. VMAT is a radiation technique combining dynamic photon fluence modulation using multi-leaf collimation (MLC) with gantry rotation to deliver a highly conformal dose distribution with improved target coverage and sparing of organs at risk (OARs).

SUMMARY:
Single institution study of safety of linac based VMAT TBI for myeloablative treatment in hematologic malignancies.

DETAILED DESCRIPTION:
Total Body Irradiation (TBI) continues to play an important role in myeloablative and non-myeloablative conditioning regimens for Allogeneic Stem Cell Transplant (ASCT). When TBI is used as part of a myeloablative regimen, it is combined with chemotherapy to eradicate malignant cells, as well as to immunosuppress the host to prevent rejection of donor hematopoietic progenitor cells (HPC).

This study is a single-institution study to assess the safety of linac based VMAT TBI for myeablative sreatment in hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patients undergoing related, unrelated (including cord blood) hematopoietic progenitor cell (HPC) transplant, in which the protocol requires >12 Gray of TBI, as part of the conditioning regimen.

   a. Conditioning regimens outlined per BMT SOP: CLNTX007: Selection of Conditioning Regimens for Blood and Marrow Transplantation - ADULTS.
3. Referral from the blood and marrow transplant (BMT) program for full-dose TBI, who meet inclusion and exclusion criterial per BMT SOPs.

   1. BMT program will initiate referral, utilizing Form: 170102, Radiation Oncology Consultation.
   2. Patients undergo pre-transplant testing, as defined in BMT SOPs:CLNAL002: Related (MRD, Haplo) Allogeneic Recipient Evaluation and Management or CLNAL011: Unrelated (MUD, MMUD, CBU) Allogeneic Recipient Evaluation and Management, per below.

   i. BMT SOP's include baseline pulmonary function tests (PFTs). Patient with decreased FVC, FEV1 and or DLCO (adjusted for hemoglobin) or pulmonary history will have pulmonary consult, at the discretion of the BMT physician prior to undergoing myeloablative radiation.

ii. Medical history and physical by BMT provider.

iii. The following laboratory tests (additional testing may be required for positive results):

* ABO group and Rh type
* Red Blood Cell Antibody Screen.
* HLA typing and confirmatory typing
* HLA antibody screen, class I and II, performed within 30 days of transplant.
* Complete blood count (CBC) with differential.
* Basic metabolic panel, including glucose and to include at a minimum electrolyte evaluation of potassium, calcium, magnesium, and phosphorus.
* Blood urea nitrogen (BUN)
* Creatinine
* Liver Function Tests including: Total bilirubin, Alkaline phosphatase, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Lactate dehydrogenase (LDH), Albumin, Total Protein, Urinalysis

Exclusion Criteria:

1. Patient receiving less than 1200 cGy of TBI
2. Previous history of thoracic radiation therapy including previous TBI
3. All premenopausal women will require a urine qualitative pregnancy test to exclude pregnancy. Pregnant women will be excluded from the study.
4. Prisoners
5. Patient not meeting transplant criteria per BMT physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve excellent coverage while sparing the lung | Up to 1 year post-transplant
  Excellent coverage while sparing the lung is quantified by meeting the following dosimetric parameters (all parameters must be met):
  1. V100%= >90% (90% of PTV volume getting 100% of the dose).
  2. D98>85% (98% of the volume getting at least 85% of the dose).
  3. Mean Lung dose <900cGy.

SECONDARY OUTCOMES:
Cumulative incidence rate of idiopathic pneumonia syndrome | Up to 100 days post-transplant
  Non-infectious pneumonia syndrome is defined by the American Thoracic Society as at least 1 of the following without concurrent infection detected on blood culture, broncoalveolar lavage, lung biopsy or sputum:
  1. There must also be the absence of cardiac dysfunction, acute renal failure, or iatrogenic fluid overload as etiology for pulmonary dysfunctionMultilobar infiltrates on chest radiograph or computed tomography (CT);
  2. Symptoms and signs of pneumonia including dyspnea, cough, cyanosis, hypoxia or pyrexia;
  3. New or increased restrictive patters on pulmonary function testing or increased alveolar to arterial oxygen difference
Occurrence of acute GVHD, transplant related mortality, or mortality in the first 100 days following transplant | 100 days post-transplant
Event Free Survival (EFS) | Up to 1 year post-transplant
Proportion of patients who achieved a mean dose to each kidney (Dmean) < 11Gy | Up to 150 days post-transplant
Proportion of patients who have achieved a maximum dose to 2cc of the entire body (D2cc) < 130% of Rx dose. | Up to 150 days post-transplant
Proportion of patients who have achieved a maximum dose to 0.03cc of OARs < 120% of Rx dose. | Up to 150 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Naamit Gerber, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to naamit.gerber@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.